CLINICAL TRIAL: NCT00901446
Title: Simultaneous Acquisition of Intravascular Ultrasound and Near Infrared Spectroscopy Data in the Coronary Artery Study
Brief Title: Study of Near Infrared Spectroscopy (NIRS) and Intravascular Ultrasound (IVUS) Combination Coronary Catheter
Acronym: SAVOIR
Status: Completed | Type: Observational
Sponsor: Infraredx (Industry)
Responsible Party: Vice President of Clinical & Regulatory Affairs, InfraReDx Inc.
Other Study IDs: 0112
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Atherosclerosis; Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Myocardial Ischemia; Myocardial Infarction | interventions — Spectrum Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Imaging: Subjects who receive intracoronary imaging with the investigative device.
  Interventions: Device: Intravascular ultrasound and spectroscopy

INTERVENTIONS:
Device: Intravascular ultrasound and spectroscopy — Intracoronary imaging with a catheter based ultrasound transducer and near infrared spectroscopy tip that is pulled back at an automated rate of 0.5 millimeters per second.
  Other Names: InfraReDx

SUMMARY:
This study is designed to evaluate the technical performance and clinical handling of a coronary catheter that includes two imaging techniques. The catheter being evaluated performs near infrared spectroscopy and ultrasound imaging of the coronary arteries. Near infrared spectroscopy is used to identify lipid or cholesterol deposits in the vessel wall and the ultrasound component provides structural information about the vessel. Combining multiple imaging techniques into a single catheter can reduce the total number of catheters required during treatment and the overall duration of cardiac catheterization. Both of these results may lead to safer procedures.

ELIGIBILITY:
Inclusion Criteria:

* >=18yrs of age.
* diagnosed with stable angina pectoris or documented silent ischemia
* scheduled for elective, non-emergent cardiac catheterization
* able to read, understand, and provide written informed consent
* >=1 obstructive stenosis (>50%DS by visual estimate)in a major native coronary artery
* clinically indicated treatment plan includes placement of a guidewire into the target artery.
* target artery has a >=30mm segment with a reference vessel diameter >=2.5mm
* target artery has a >50%DS luminal narrowing

Exclusion Criteria:

* Subject unwilling or unable to provide written informed consent.
* Subject unwilling to comply with protocol
* Subject is pregnant
* Subject is of childbearing potential without negative pregnancy test.
* Subject received prolonged CPR within 2 weeks of enrollment procedure
* Subject is intubated.
* Subject is diagnosed with an acute coronary syndrome.
* Subject has severe persistent hypertension.
* Subject has renal dysfunction or insufficiency.
* Subject has an abnormal platelet count.
* Subject has low hemoglobin levels.
* Subject has active liver disease or dysfunction.
* subject diagnosed with acute pulmonary edema or congestive heart failure.
* Subject diagnosed or suspected to have acute myo-, peri-, or endo- carditis, cardiac tamponade, or dissected aortic aneurysm.
* Subject has significant valvular heart disease, cardiomyopathy, or congenital heart disease.
* Subject has history of intracranial bleeding or aneurysm.
* Subject has a history of stroke that precludes the use of routine antithrombotic agents during PCI?
* Subject has known hypercoagulable state, coagulopathy, or abnormal bleeding.
* subject has family history of coagulopathy or bleeding diathesis.
* subject has undergone PCI in the last 30days.
* subject enrolled or participating in pharmaceutical study in last 30 days.
* subject enrolled or participating in medical device treatment study in last 30 days.
* subject has obstructive LMCA disease.
* subject has multivessel CAD that requires additional treatment in a separate procedure with 30days of enrollment.
* subject has unprotected left main disease.
* three vessel intervention is required during enrollment procedure.
* target artery is the left circumflex artery.
* target artery is accessed through a vein or arterial graft.
* target artery is tortuous
* target artery contains segments of severe calcification
* target artery has >2 serial obstructions exceeding 50%DS.
* target artery has an aneurysm or suspected aneurysm.
* target artery has <=1 TIMI flow.
* target lesion is >99% DS.
* target lesion is severely calcified
* target lesion has angiographic characteristics of thrombus.
* target lesion has angiographic characteristics of ulceration.
* target lesion has inclusion of a side branch greater than 1mm.
* target lesion is located in a vessel segment with >4.0mm reference vessel diameter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the patients presenting to the cardiac catheterization laboratory for elective cardiac catheterization.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Obtain registered NIRS and IVUS data from a single catheter placement and single imaging run. | day 0

SECONDARY OUTCOMES:
The imaging tip can be positioned in the mid segment of the target artery. | day 0
The lumen boundary of the target stenosis can be distinguished within the IVUS data set. | day 0
The external elastic membrane (EEM) of the target stenosis can be distinguished within the IVUS data set. | day 0
The lumen and EEM can be distinguished in the same cross section of the IVUS data set. | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Serruys, MD, Principal Investigator — Erasmus Medical Centre
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

REFERENCES:
- See also: Sponsor Website — http://www.infraredx.com